CLINICAL TRIAL: NCT01029509
Title: An Open-label, Non-randomized Study to Assess the Pharmacokinetics, Dose Limiting Toxicity and Maximum Tolerated Dose of OPB-31121 in Subjects With Advanced Leukemias or Myelodysplastic Syndromes
Brief Title: Study to Assess OPB-31121 in Advanced Leukemias or Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Colloborator-Sponsor decision to terminate.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0488
Record Dates: First submitted 2009-12-08; First posted 2009-12-10 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: Advanced Leukemia; Acute myeloid leukemia; ALL; Chronic myeloid leukemia blast crisis; CMS; Acute lymphocytic leukemia; Chronic lymphocytic leukemia; Myelodysplastic syndromes; MDS; OPB 31121
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-31121 (Experimental): OPB-31121 200 mg twice daily for 21 days followed by 7 days of rest
  Interventions: Drug: OPB 31121

INTERVENTIONS:
Drug: OPB 31121 — Starting dose of 200 mg (two 100 mg tablets) twice a day for 21 days followed by 7 days of rest.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of OPB-31121 that can be given to patients with leukemia or myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
The Study Drug:

In studies that have been performed in animals, OPB-31121 has been shown to stop certain changes to proteins in the body. Stopping these changes may have an effect on tumor cells. How OPB-31121 works is not fully known.

Study Groups:

The first 3 participants enrolled in the study will receive the lowest level of OPB-31121. Each additional group of 3 or 4 participants will receive a dose level dependent upon how the previous group responded to the study drug.

You may have up to 13 study "cycles" (about 273 days). During each 28 day study cycle, you will receive the study drug for 21 days and then "rest" (no study drug) for 7 days. The cycle is 28 days, 21 days of drug, 7 days of rest.

Study Drug Administration:

The study drug is a pill that should be taken at the same time each day. You should drink 8 ounces (1 cup) of room temperature, non-carbonated water when you take the study drug.

You will eat a snack or meal within 30 minutes after taking the study drug. You should remain sitting upright or standing for at least 30 minutes after taking the drug.

Study Visits for AML, ALL, or MDS participants:

On Day 1 of Cycle 1, you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Urine will be collected for routine tests.
* Women who are able to have children will have a urine pregnancy test.
* Blood (about 6 tablespoons total) will be drawn about 10 times. These blood draws will be for routine tests, heart, thyroid testing, pharmacokinetic (PK) testing, and genotyping. PK testing measures the amount of study drug in the body at different time points. Genotyping tests are tests that look at pieces of your DNA called genes. These tests will look at some specific genes that may predict how your body may break down certain types of drugs. A small needle called a "heparin lock" may be inserted into a vein to make these multiple blood draws easier.

On Day 2 of Cycle 1, blood (about 2 tablespoons) will be drawn for heart, PK, and biomarker testing.

On Days 8, 15 and 21 of Cycle 1:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Urine will be collected for routine tests.
* Blood (about 2 tablespoons) will be drawn for routine, heart, and thyroid testing.
* Blood (about 6 tablespoons total) will also be drawn for PK testing. Blood will be drawn a total of 10 times, with the last blood draw about 10 hours after you receive the study drug.
* Blood (about 1/2 tablespoon) will be drawn for biomarker testing (Day 21 only).

On Day 22 of Cycle 1, blood (about 1 tablespoon each time) will be drawn 2 times for PK testing.

On Day 23 of Cycle 1, blood (about 1 tablespoon) will be drawn 1 time for PK testing.

On Day 28 of Cycle 1, you will have the following procedures performed:

* You will have an ECG.
* You will have a physical exam, including measurement of your vital signs.
* You will have a bone marrow aspiration sample taken to check the status of the disease. This sample will be taken after you have taken the study drug and only at the end of each odd cycle.

On Day 1 of Cycles 2-13, you will have the following tests and procedures will be performed:

* Blood (about 1-1/2 tablespoons) and urine will be collected for routine, heart, and thyroid tests.
* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Women who are able to have children will have a urine pregnancy test.
* On Day 1 of Cycles 2 and 3 only, blood (less than 1 tablespoon) will be drawn for biomarker tests.
* You will have a MUGA scan.
* If your doctor thinks it is needed, you will have a bone marrow aspiration/biopsy.

Study Visits for CLL or CML participants:

On Day 1 of Cycle 1, you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Urine will be collected for routine tests.
* Blood (about 8 tablespoons total) will also be drawn a total of 10 times for routine, heart, thyroid, biomarker, genotyping, and PK testing. The last blood draw will be 24 hours after you receive the study drug (Day 2). A small needle called a "heparin lock" may be inserted into a vein to make these multiple blood draws easier.
* Women who are able to have children will have a urine pregnancy test.
* If your doctor thinks it is needed, you will have a bone marrow biopsy.

On Day 2 of Cycle 1, blood (about 2 tablespoons) will be drawn 24 hours after your study drug dose for heart and PK testing.

On Days 8 and 15 of Cycle 1, blood (about 7 tablespoons) will be drawn for routine and PK testing.

On Days 21 of Cycle 1, you will have an ECG. Blood (about 8 tablespoons in total) will be drawn about 8 times for PK, routine, heart, thyroid, and biomarker testing.

On Days 22 of Cycle 1, blood (about 1 tablespoon each time) will be drawn 2 times for PK testing.

On Day 23 of Cycle 1, blood (about 1 tablespoon) will be drawn 1 time for PK testing.

During Cycles 2-13, blood (about 1 tablespoon) will be drawn every 2 weeks for routine, heart, and thyroid testing.

On Day 1 of Cycles 2-13, you will have the following tests and procedures performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG and MUGA scan.
* Blood (about 2 tablespoons) will be drawn for routine, heart, thyroid, and biomarker tests.
* Women who are able to have children will have a urine pregnancy test.
* During Cycles 2-3 only, blood (about 1 tablespoon) will be drawn for biomarker testing.

End-of-Study Visit:

Once you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Blood (about 7 tablespoons) will be drawn for routine, heart, thyroid, and PK tests.
* Urine will be collected for routine tests.
* If you have AML, ALL or MDS, blood (about 1-1/2 tablespoons) will be drawn for biomarker testing.

Follow Up:

Your doctor or other study staff will call you about 30 days after your final visit to see how you have been feeling. The phone call will take about 5-10 minutes.

This is an investigational study. OPB-31121 is not FDA approved or commercially available. At this time, OPB-31121 is only being used in research. Up to 48 patients will take part in this multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a diagnosis of treatment resistant or relapsed AML, ALL, or CLL for whom no standard treatment therapies are expected to result in durable remission. Subjects with advanced MDS should have failed lenalidomide or a hypomethylating agent. Subjects with CLL should have failed or relapsed after prior fludarabine and Campath. Subjects with CML should have previously exhausted standard therapy which provides clinical benefit. In addition, untreated subjects not eligible for standard therapy or unwilling to receive standard therapy with the above diagnosis will be eligible.
2. Male and female subjects > / = 18 years of age
3. Male and female subjects who are surgically sterile (ie, have undergone orchidectomy or hysterectomy, respectively); female subjects who have been postmenopausal for at least 24 consecutive months; or male and female subjects who agree to remain abstinent or to begin two acceptable methods of birth control from one week prior to drug administration through 30 days (for females) and 90 days (for males) from the last dose of study medication.
4. (continued from #3) If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device (IUD), condom, diaphragm, cervical cap or sponge with spermicide.
5. Adequate liver function defined as </= 2.5 * institutional upper limit of normal (ULN), </= 2.5 * institutional ULN for alanine transaminase (ALT), aspartate transaminase, (AST) and bilirubin within normal limits unless Gilbert disease has been documented. .
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. In the absence of rapidly proliferative disease, a minimum of 2 weeks should elapse since prior standard or experimental therapy. Subjects must have recovered to grade less than or equal to 1 from any prior nonhematologic toxicities associated with any previous treatments. Use of leukopheresis or hydrea up to 48 hrs prior to the start of the study will be allowed in presence of proliferative disease. Use of hydrea will be permitted up to 5 days in each cycle for the control of proliferative disease.
8. All eligible subjects must have received prior therapy (including chemotherapy, radiation therapy or surgery) greater than or equal to 2 weeks prior to study entry (Screening) and have recovered to Grade 1 toxicity from any prior non-hematological toxicity and to Grade 2 toxicity from any prior hematological toxicity except for thrombocytopenia defined as Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding following investigator's assessment of causality and positive relationship to study medication before participation in this trial.
9. For CLL subjects only, all subjects with Rai Stages III-IV are eligible. For subjects with Rai stage 0-I disease, one or more indications for treatment as defined by the NCI sponsored Working Group must exist: • Massive or progressive splenomegaly; OR • Massive lymph nodes; nodal clusters, or progressive lymphadenopathy; OR • Grade 2 or 3 fatigue; or fever > / = 100.5° F or night sweats for greater than 2 weeks without documented infection; or presence of weight loss > / = 10% over the preceding 6 months;
10. (continued from #9) OR • Progressive lymphocytosis with an increase in lymphocyte count of > / = 50% over a 2- month period or an anticipated doubling time of less than 6 months.
11. For CML, subjects who have exhausted standard therapy which provides clinical benefit.
12. Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the study.
13. Subjects must have a life expectancy of > 3 months.
14. Subjects must have a normal ejection fraction (>/= 50%) as measured by multiple gated acquisition (MUGA) scan.
15. Subjects must have a normal serum creatinine (at baseline only) with a measured 24 hour creatinine clearance of > 60 cc/min.

Exclusion Criteria:

1. Clinically significant condition in past medical history, or at the screening physical examination, that in the investigator's or sponsor's opinion may place the subject at risk or interfere with outcome variables.
2. Subjects with active central nervous system (CNS) involvement by leukemia. Subjects with prior history of CNS disease will qualify if active disease is ruled out by imaging studies or spinal tap
3. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
4. Subjects having taken an investigational drug or therapy within 14 days prior to dosing.
5. Subjects who are pregnant or breast feeding. A negative serum pregnancy test must be confirmed prior to the first dose of study medication for WOCBP.
6. Use of CYP3A4-enzyme inhibiting drugs and food; use of CYP3A4-enzyme inducing drugs and food; use of CYP2C9-enzyme inhibiting drugs; and use of CYP2C9 enzyme inducing drugs. Others: propranolol, lidocaine, propafenone, verapamil, nitroglycerin, and midazolam.
7. Subjects with history of coagulopathy (or taking anticoagulants) including deep vein thrombosis (DVT)/ PE, unstable angina, myocardial infarction and stroke within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Assessed at end of 28 day cycle for each dose cohort
  MTD defined as highest dose level at which < 2 of 6 subjects experience dose limiting toxicity (DLT) during the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org